CLINICAL TRIAL: NCT01672801
Title: Using Nimodipine, a Calcium Channel Blocker, to Prevent LH Surge in Women Undergoing Controlled Ovarian Stimulation and Intrauterine Insemination: a Double-blinded, Randomized Controlled Study
Brief Title: Nimodipine to Prevent LH Surge During Ovulation Induction: Blinded Placebo-controlled RCT
Acronym: NIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston IVF (Other)
Collaborators: Village Fertility Pharmacy (Industry)
Responsible Party: Principal Investigator, Alan Penzias, Associate Professor of Obstetrics, Gynecology and Reproductive Biology, Boston IVF
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012P-000186
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Unexplained Infertility; Polycystic Ovarian Syndrome; Anovulatory
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation | interventions — Nimodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): All subjects in both arms will receive Clomid 100 mg tablets by mouth for 5 days prior to receiving either placebo comparator or active comparator. Placebo comparator subjects will receive 8 total doses of liquid placebo orally 4 times a day for 8 total doses in pre-filled liquid placebo containing syringes
  Interventions: Drug: Placebo
- Nimodipine (Active Comparator): All subjects in both arms will receive Clomid 100 mg tablets by mouth for 5 days prior to receiving either placebo comparator or active comparator. Active comparator subjects will receive Nimodipine 30mg liquid orally 4 times a day for 8 total doses in pre-filled syringes
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Placebo — oral administration
  Arms: Placebo
Drug: Nimodipine — oral administration
  Other Names: Nimotop
  Arms: Nimodipine

SUMMARY:
The main purpose of this study is to test the effectiveness of nimodipine in preventing a luteinizing hormone (LH) surge in women undergoing ovulation induction with clomiphene citrate. It is important to prevent the premature LH surge in controlled ovarian stimulation to allow adequate recruitment of follicles, proper maturation of a dominant follicle before ovulation, and effectively time insemination with semen to allow fertilization of a mature egg to occur.

The investigators are also conducting this study to determine medication side effect profile (including lightheadedness or dizziness from low blood pressure or rapid heart rate, headache, and nausea), patient treatment compliance, and clinical pregnancy (positive pregnancy test and ultrasound evidence of fetal heart rate). Finally, LH and follicle stimulating hormone (FSH) serum levels will be measured to determine effect of nimodipine on these hormones.

As a calcium channel blocker, nimodipine has been shown to block calcium mediated release of gonadotropin releasing hormone in animal and preliminary human studies. The investigators hypothesize that nimodipine, a calcium channel blocker, will prevent or delay the LH surge during controlled ovarian stimulation cycles using clomiphene citrate in subfertile patients undergoing assisted reproduction with intrauterine insemination (IUI).

DETAILED DESCRIPTION:
After enrollment, subjects will be randomized to Placebo Comparator or Active Comparator. All subjects will receive Clomid 100 mg for 5 days for the purpose of ovarian follicle recruitment. Intervention will be initiated once ovarian follicle maturation has been documented (≥1 ovarian follicle size of ≥ 17mm) and the absence of a premature LH surge has been confirmed - this will be classified as intervention day 0. Subjects will receive their assigned comparator (Placebo or Active) according the schedule below:

* Intervention Day 0 - noon / afternoon / bedtime (3 doses)
* Intervention Day 1 - morning / noon / afternoon / bedtime (4 doses)
* Intervention Day 2 - morning (1 dose) Serum hormone levels and ultrasound examination will occur on days 0,1 and 2 for all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-40 years at the time of enrollment
* Both ovaries intact by history and ultrasound assessment
* Early follicular phase (day 2-4) serum FSH level <20 mIU/mL
* Diagnosis of subfertility with a recommended treatment of COH and IUI
* Providing written informed consent in English

Exclusion Criteria:

* Body mass index (BMI) >38 kg/m2
* Early follicular phase (day 2-4) serum FSH level ≥20 mIU/mL
* History of overstimulated cycle defined as >3 mature follicles of ≥17 mm
* Abnormal uterine cavity and/or tubal disease (as evidenced by sonohysterogram or hysterosalpingogram)
* Diagnosis of infertility with a clear indication for in-vitro fertilization, such as bilateral tubal occlusion
* Severe male factor infertility: Total Motile Sperm Count < 2x106 post washing (sperm deemed inadequate for IUI preparation)
* Any ovarian or abdominal abnormality that may interfere with adequate TV ultrasound evaluation
* Absence of one or both ovaries
* Any contraindication to being pregnant or carrying a pregnancy to term
* Unexplained gynecological bleeding
* Any medical condition that would jeopardize the patient or the integrity of the data obtained including:
* Prior reaction or side effects from previous calcium channel blocker use
* Any medical condition that may interfere with the absorption, distribution, metabolism or excretion of nimodipine such as hepatic disease, hypertension, seizure, concurrent infection, depression, reflux (see #12 below).
* Mental health status resulting in cognitive or emotional impairment that would preclude study participation
* The concurrent use of any of the following drugs: [These medications have been shown to effect the availability of the medication or worsen hypotension symptoms]
* Antihypertensives (eg. ACE inhibitors, alpha-adrenergic blocking agents,methyldopa, beta-blockers, diuretics, PDE5 inhibitors, and other calcium antagonists)
* Antiepileptics (eg. phenobarbital, phenytoin, carbamazepine or valproic acid)
* Macrolide antibiotics (eg, erythromycin)
* Azole antimycotics (eg, ketoconazole)
* HIV protease inhibitors (eg, ritonavir)
* Antidepressants (eg, nefazodone and fluoxetine)
* Cimetidine
* Patient unable to communicate adequately with the investigators and to comply with the requirements of the study
* Unwillingness to give written informed consent

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan S Penzias, MD, Principal Investigator — Beth Israel Deaconess Medical Center / Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen EC, Javors MA, Norris C, Siler-Khodr T, Schenken RS, King TS. Dependence of 3',5'-cyclic adenosine monophosphate--stimulated gonadotropin-releasing hormone release on intracellular calcium levels and L-type calcium channels in superfused GT1-7 neurons. J Soc Gynecol Investig. 2004 Sep;11(6):393-8. doi: 10.1016/j.jsgi.2004.02.010. PMID 15350253
- [Background] Krsmanovic LZ, Stojilkovic SS, Merelli F, Dufour SM, Virmani MA, Catt KJ. Calcium signaling and episodic secretion of gonadotropin-releasing hormone in hypothalamic neurons. Proc Natl Acad Sci U S A. 1992 Sep 15;89(18):8462-6. doi: 10.1073/pnas.89.18.8462. PMID 1326758
- [Background] Nunez L, Villalobos C, Boockfor FR, Frawley LS. The relationship between pulsatile secretion and calcium dynamics in single, living gonadotropin-releasing hormone neurons. Endocrinology. 2000 Jun;141(6):2012-7. doi: 10.1210/endo.141.6.7491. PMID 10830284

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Nimodipine
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — Screen Failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nimodipine | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Full Range); unit: years] | 33 [31 to 36] | 37 [31 to 42] | 35 [31 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: LH Surge
Description: Compare the change between placebo treated and nimodipine treated patients by the presence or absence of an LH surge on intervention Day 1 and Day 2. LH surge will be determined by serum LH levels at least two times the baseline serum LH (baseline serum LH = (cycle day 3 serum [LH] + cycle day 7 serum [LH])/2).
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nimodipine
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

2. Secondary Outcome: Number of Participants Experiencing Side Effects
Description: Medication side effect profile including: symptomatic hypotension (Note: vital signs will be recorded), symptomatic tachycardia (Note: vital signs will be recorded), headache, nausea. These will be self-reported with constructed questionnaire.
Time Frame: Starting day 0 of intervention to pregnancy test (approximately 15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nimodipine
Number analyzed (Participants) | 9 | 9
Participants | 3 | 4

3. Other Pre Specified Outcome: Gonadotropin Levels
Description: Calculated changes in serum LH, FSH, and estradiol levels between patients in nimodipine and placebo arms
Time Frame: Intervention day 0 to ovulation (approximately 1-7 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo | Nimodipine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 4/9
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Nimodipine (N=9)
headache (General disorders) | 2 (2) | 3 (3)
Dizziness (General disorders) | 0 (0) | 3 (3)
Acne (General disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes